CLINICAL TRIAL: NCT01972711
Title: A Randomized, Double-blind, Placebo-controlled, Single-dose, Study of the Effects of SEP 363856 and Amisulpride on BOLD-fMRI Signal in Healthy Male and Female Volunteers With High or Low Schizotype Characteristics.
Brief Title: Study Assessing SEP-363856 in Male and Female Volunteers With High or Low Schizotype Characteristics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-104
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856; Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SEP-363856 (Experimental): Single-dose SEP-363856 50 mg
  Interventions: Drug: SEP-363856
- Amisulpride (Active Comparator): Single-dose Amisulpride 400 mg.
  Interventions: Drug: Amisulpride
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-363856 — SEP-36385625 as a single oral dose of 50 mg
  Arms: SEP-363856
Drug: Amisulpride — Amisulpride as a single oral dose of 400 mg
  Arms: Amisulpride
Drug: Placebo — single oral dose placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the effects of a single dose of SEP-363856 in healthy male and female volunteers with high or low schizotype characteristics.

DETAILED DESCRIPTION:
The study is a randomized, double-blind, placebo-controlled functional magnetic resonance imaging (fMRI) study of the effects of a single dose of SEP-363856 and amisulpride on blood oxygen level dependent (BOLD) signal in healthy male and female volunteers with high or low schizotype characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 45 years, inclusive, at Day 1.
* Subject must be healthy as determined by the Investigator, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring within four weeks of randomisation. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Subject must be normotensive with sitting (5 minutes) blood pressure between the range of 90 to 150 mm Hg systolic, inclusive, and 60 to 90 mm Hg diastolic, inclusive, at Screening.
* Subject must have sitting (5 minutes) heart rate ≥ 50 beats per minute at Screening.
* Subject must agree to use one of the following birth control/contraception methods from Screening until 90 days after receiving study drug.
* Female subject of child bearing potential (≤ 65 years) should be surgically sterile or abstinent or, if sexually active, must use an adequate method of contraception in addition to their partner(s) using a barrier method.
* Male subject with female partner(s) of childbearing potential must take appropriate precautions to avoid fathering a child and use barrier contraception, in addition to their female partner(s) using another method.
* Male subject must not donate sperm.
* Acceptable forms of contraception are as follows:
* Barrier methods: condoms, diaphragms, cervical caps; with a spermicide foam, gel, film, cream or pessary.
* Non-hormone containing intrauterine methods: intrauterine devices or systems.
* Other: prescription oral contraceptives, contraceptive injections, contraceptive implant, contraceptive vaginal ring, hormonal intrauterine device, double-barrier method, contraceptive patch, or male partner sterilisation.
* Subject must have normal ECG results, including QTcF < 450msec (for men) or < 470 ms (for women) (based on the Fridericia correction where QTcF = QT/RR0.33) at Screening.
* Subject must be a completely fluent English speaker who, in the opinion of the Investigator, is capable of completing the fMRI and behavioural tasks.
* Subject must be right-handed.
* Subject must have acceptable weight as defined by BMI (weight [kg]/height [m]²) range of 18 to 35 kg/m², inclusive at Screening.
* Subject must be a non-smoker or light smoker (≤ 10 cigarettes per day).
* Subject must have signed the informed consent form prior to the first study-related procedure indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
* Subject in the low schizotypy group must have an SPQ score < 10 at Screening.
* Subject in the high schizotypy group must have an SPQ score >43 at Screening

Exclusion Criteria:

* Subject with a history of alcohol or substance dependence within the last 12 months from Screening.
* Subject with a positive urine drug screen at Screening or Day 1. One re-test within 1 to 3 days is permitted if positive result is believed to be due to licenced opiate-based medication or ingestion of poppy seeds. In this event, re-test result will be used for assessing entry criterion and must be completed prior to randomisation.
* Subject with a positive alcohol breath test at Screening or Day 1.
* Female subject with a positive pregnancy test at Screening or Day 1.
* Female subject currently pregnant or trying to get pregnant or currently breast feeding.
* Subject who consumes large amounts of caffeinated drinks (more than 8 cups of standard caffeinated drinks (tea, instant coffee) or 6 cups of stronger coffee or other drinks containing methylxanthines such as coca cola or Red Bull per day).
* Subject with a relevant history, or presence upon clinical examination, of cardiac, ophthalmologic, pulmonary, endocrine (diabetes), blood disease, gastro-intestinal, hepatic or renal disease or other condition which in the opinion of the Investigator could interfere with the test procedures.
* Subject with a history of cancer, except for basal cell or Stage 1 squamous cell carcinoma of the skin which has been in remission for at least 5 years prior to Day 1.
* Subject meets the diagnostic criteria for schizophrenia, or any other psychotic disorder, as determined by the SCID-I at Screening
* Subject with a history of, or presents (in the opinion of the Investigator) with, significant neurological or psychiatric conditions (such as stroke, traumatic brain injury, depression, seizures, space occupying lesions, multiple sclerosis, Parkinson's disease, vascular dementia, transient ischemic attack, schizophrenia, blackouts requiring hospitalisation).
* Subject with a history of positive HIV test.
* Subject with a history of, or current condition of, migraine headaches or has undergone operations to the head.
* Subject with a significant hearing impairment which, in the opinion of the Investigator, may interfere with the performance of the behavioural tasks or fMRI tasks.
* Subject with a significant visual impairment including colour blindness, or history of ocular treatment including corrective laser eye surgery, or ongoing condition, which in the opinion of the Investigator may interfere with the performance of the behavioural tasks or fMRI tasks.
* Subject received prescribed medication within 28 days prior to Day 1 (apart from the contraceptive pill). Subjects who have taken prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety (see Section 10.2, Concomitant Medications).
* Subject received non-prescription medication, including supplements such as vitamins and herbal supplements within 48 hours prior to Day 1 (apart from paracetamol). Subjects who have taken non-prescription medication may still be entered into the study, if, in the opinion of the Investigator, the medication received will not interfere with the study procedures or compromise safety (see Section 10.2, Concomitant Medications).
* Subject received an experimental drug and / or used an experimental medical device within 30 days of randomisation or within a period less than 5 times the drug's half-life, whichever is longer.
* Subject with a known hypersensitivity to SEP-363856 or amisulpride or any of their excipients.
* Subject with a history of severe drug allergy or hypersensitivity.
* Subject who is unable or unwilling to comply with study procedures, including study prohibitions and restrictions (see Section 10.2, Concomitant Medications and Section 10.3, Restrictions).
* Subject with previous experience with the ETB.
* Subject with a diagnosis of dyslexia.
* Subject with a history of claustrophobia or inability to tolerate scanner environment.
* Subject who fulfills any of the MRI contraindications on the standard site radiography screening questionnaire (e.g. history of surgery involving metal implants).
* Subject with a clinically relevant structural brain abnormality as determined by prior MRI scan.
* Subject with planned medical treatment within the study period that might interfere with the study procedures.
* Subject who is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator.
* Subject is a staff member or the relative of a staff member, or is in a subordinate relationship with the Investigator.
* Subject answers "yes" to "Suicidal Ideation" Items 4 or 5 on the C-SSRS.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI activity in key regions of interest (ROIs) while performing the Monetary Incentive Delay (MID), N-back, and Signal detection (SD) tasks after a single-dose of study medication | Up to 6 Weeks

SECONDARY OUTCOMES:
Behavioural performance in the MID task, includes measurements of trial accuracy, trial duration, trial reaction time and amount of money won. | Up to 6 Weeks
Behavioural performance in the N-back task, includes measurements of accuracy (% correct for each trial type), reaction time and target sensitivity (d'). | Up to 6 Weeks
Behavioural performance in the SD task, includes measurements of correct and incorrect responses. | Up to 6 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Department of Psychiatry, University of Oxford, Warneford Hospital, Headington, Oxford
  - University of Manchester, Neuroscience and Psychiatry Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Perini F, Nazimek JM, Mckie S, Capitao LP, Scaife J, Pal D, Browning M, Dawson GR, Nishikawa H, Campbell U, Hopkins SC, Loebel A, Elliott R, Harmer CJ, Deakin B, Koblan KS. Effects of ulotaront on brain circuits of reward, working memory, and emotion processing in healthy volunteers with high or low schizotypy. Schizophrenia (Heidelb). 2023 Aug 7;9(1):49. doi: 10.1038/s41537-023-00385-6. PMID 37550314